CLINICAL TRIAL: NCT04569435
Title: Phase 2a Safety, Tolerability, Pharmacokinetic (PK), and Pharmacodynamic (PD) Study of Intravenous ANX005 in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Study of ANX005 in Adults With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANX005-ALS-01
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANX005 (Experimental): Participants will receive induction dosing of ANX005 on Days 1 and 5 or 6, followed by maintenance doses of ANX005 every 2 weeks up to Week 22.
  Interventions: Drug: ANX005

INTERVENTIONS:
Drug: ANX005 — IV Infusion

SUMMARY:
This study is a multi-center, open-label study of intravenous (IV) ANX005 in participants with ALS.

DETAILED DESCRIPTION:
In this Phase 2a, multi-center, open label, proof-of-biology study, ANX005 will be administered to participants with ALS.

The study consists of approximately 22 weeks of treatment and approximately 14 weeks of follow-up. All participants will be contacted by phone 6 months after study completion.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of ALS according to the World Federation of Neurology revised EI Escorial criteria.
* Onset of weakness within 3 years prior to Day 1 visit.
* Slow Vital Capacity ≥ 50% of predicted normal adjusted for sex, age, and height (from the sitting position).
* ALS Functional Rating Scale-Revised (ALSFRS-R) ≥ 30 at the Screening visit (Week -2).
* If female, must be postmenopausal, surgically sterilized, or childbearing potential must agree to use highly effective methods of contraception from Screening until 3 months after the last infusion with study medication.
* Males with a woman partner of childbearing potential must agree to use highly effective methods of contraception from Screening until Week until 3 months after the last infusion with study medication.
* Documented history of vaccinations within 5 years prior to Screening visit against encapsulated bacterial pathogens or willing to undergo vaccinations.

Key Exclusion Criteria:

* Clinically significant intercurrent illness, medical condition, or medical history that would jeopardize the safety of the participant, limit participation, or compromise the interpretation of the data derived from the participant.
* Participants with body weight > 150 kilograms.
* Antinuclear antibodies (ANA) titer ≥ 1:160 (for either of the 2 ANA results a minimum of 2 weeks apart) during the Screening Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Treatment-Emergent Adverse Events | Up to Week 36

SECONDARY OUTCOMES:
Serum Concentrations of ANX005 | Up to Week 36
Maximum Observed Serum Concentration (Cmax) of ANX005 | Up to Week 36
Area Under the ANX005 Serum Concentration-Time Curve | Day 1 and Week 22
Change from Baseline in Free Complement (C) 1q Serum Concentrations | Baseline, up to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hoehn, MD, PhD, Study Director — Annexon, Inc.
Locations (8):
- United States (4):
  - Annexon Investigational Site 04, Phoenix, Arizona
  - Annexon Investigational Site 01, Orange, California
  - Annexon Investigational Site 02, Gainesville, Florida
  - Annexon Investigational Site 03, Tampa, Florida
- Canada (4):
  - Annexon Investigational Site 10, Edmonton, Alberta
  - Annexon Investigational Site 09, Toronto, Ontario
  - Annexon Investigational Site 07, Montreal, Quebec
  - Annexon Investigational Site 08, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No